CLINICAL TRIAL: NCT02130596
Title: A Pilot Study of an Acceptance-Based Behavioral Intervention Versus Nutritional Counseling for Weight Loss in Psychotic Illness
Brief Title: An Acceptance-Based Behavioral Intervention vs. Nutritional Counselling for Weight Loss in Psychotic Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Rohan Ganguli, Senior Scientist, Canada Research Chair, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 132/2013
Record Dates: First submitted 2014-05-01; First posted 2014-05-05 (Estimated); Last update posted 2014-11-07 (Estimated); Status verified 2014-11

CONDITIONS: Psychotic Illnesses

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acceptance-Based Behavioral Intervention (Experimental)
  Interventions: Behavioral: Acceptance-Based Behavioral Intervention
- Nutritional Counselling (Active Comparator)
  Interventions: Other: Nutritional Counselling

INTERVENTIONS:
Behavioral: Acceptance-Based Behavioral Intervention
  Arms: Acceptance-Based Behavioral Intervention
Other: Nutritional Counselling
  Arms: Nutritional Counselling

SUMMARY:
Obesity occurs at 2-3 times the general population rate in persons living with a psychotic illness. The risk of obesity-related serious medical conditions like diabetes and heart disease are also two to three times higher in this population. Traditional behavioral weight management approaches help more than half of these individuals to lose weight, but a significant proportion are not helped. This pilot study is intended to determine the feasibility, efficacy, acceptability, and potential clinical utility of an intervention that integrates mindfulness, acceptance, distress tolerance, and motivation and commitment combined with traditional behavioral strategies for weight loss. This is the first study to investigate such an acceptance-based behavioral intervention for weight loss in psychotic illness. The results from this study will help to determine whether future research in this area is warranted with a larger sample, over a longer period of time.

Primary hypothesis: Weight loss will be greater in individuals who receive the acceptance based behavioral intervention, relative to those who receive nutritional counseling.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 25.0
* Diagnosed psychotic illness (i.e., schizophrenia, schizoaffective disorder, schizophreniform disorder, bipolar I disorder, major depressive disorder with psychotic features, substance-induced psychotic disorder, and psychotic disorder not otherwise specified).

Exclusion Criteria:

* Inability to provide informed consent
* Prediabetes or type 2 diabetes mellitus
* Current enrollment in another formal weight management program
* Brief Psychiatric Rating Scale (BPRS) ratings of 4 or more on any one of Grandiosity (Item #6), Suspiciousness (Item #7), Hallucinations (Item #8), Unusual Thought Content (Item #9), or Conceptual Disorganization (Item #10), or a BPRS total score of 80 or more.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-02; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Weight (kg) | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rohan Ganguli, M.D., Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada